CLINICAL TRIAL: NCT05731206
Title: Study to Assess Hypoallergenicity of a Hydrolysed Protein Formula in Children With Confirmed Cow's Milk Allergy
Brief Title: Hypoallergenicity of a Hydrolyzed Protein Infant Formula
Acronym: HYPO STORY
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal discussions
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SBB22R&40330
Record Dates: First submitted 2022-12-23; First posted 2023-02-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Cow's Milk Allergy
Keywords: Infant formula; Hypoallergenicity
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Crossover assignment and an observational, single-arm, follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrolized protein formula (Experimental): hydrolysed protein formula
  Interventions: Other: Hydrolyzed protein infant formula
- Control formula (Placebo Comparator): commercially available hypoallergenic infant formula
  Interventions: Other: commercially available hypoallergenic infant formula

INTERVENTIONS:
Other: Hydrolyzed protein infant formula — Hydrolyzed protein infant formula
  Arms: hydrolized protein formula
Other: commercially available hypoallergenic infant formula — commercially available hypoallergenic infant formula
  Arms: Control formula

SUMMARY:
Study to demonstrate hypoallergenicity of a hydrolysed protein infant formula in a population of children with confirmed cow's milk allergy.

DETAILED DESCRIPTION:
The study consists of a double-blind, placebo-controlled food challenge, followed by a single arm open challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children aged up to 3 years.
2. Diagnosed with cow's milk allergy (or re-confirmed), within two months prior to the study (challenge day #1), by:

   1. Physician-supervised double-blind oral food challenge; or
   2. Physician-supervised open oral food challenge that elicited objective immediate allergic reactions; or
   3. Report of convincing allergic reaction to cow's milk or a milk-containing food product, in conjunction with presence of milk-specific serum Immunoglobuline E (IgE) level > 0.7 kilounit per liter (U/L) or by skin prick test (wheal size ≥ 3mm).
3. Willing to switch to a different hypoallergenic formula
4. On elimination diet (commercially available, hypoallergenic infant formula ) and free of clinical symptoms, or with controlled stable symptoms, for at least one week preceding the study (challenge day #1).
5. Expected minimal consumption of 144ml of test product/day during the open challenge.
6. Written informed consent provided by parents/guardians, according to local law.

Exclusion Criteria:

1. Infants/children who are more suitable to use AAF as first-line formula, including but not limited to those with high risk of anaphylaxis (prior history of anaphylaxis and currently not using eHF) or severe forms of non-IgE-mediated CMA such as eosinophilic oesophagitis, enteropathies, or Food Protein-Induced Enterocolitis Syndrome (FPIES).
2. Diagnosis or known allergy to any of the ingredients in the test product.
3. Congenital anomalies which will interfere with oral feeding or gastrointestinal tract, other chronic diseases (including but not limited to cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, immunological and endocrine disease), major gastrointestinal disease/abnormalities, or any other medical condition that could interfere with the identification of allergic reactions.
4. (Twin / triplet) sibling of an infant/child already participating in the study.
5. Investigator's uncertainty about the willingness or ability of the subject and his/her parents to comply with the protocol requirements.
6. Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.
7. Employees and/or children/family members or relatives of employees of Nutricia Research or the participating study sites.

Ages: 0 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Hypoallergenicity | 25-35 days
  The percentage of children tolerating the formula tested by double-blind, placebo-controlled food challenge and a subsequent open challenge.

OTHER OUTCOMES:
Relevant parameters routinely collected in the clinic | 25-35 days
  e.g serum IgE results
Incidence, seriousness, severity and relatedness of Adverse Events | 25-35 days
  Safety and tolerance parameters
Demographics characteristics | at baseline
  Demographics characteristics
Relevant parameters routinely collected in the clinic | 25-35 days
  e.g. skin prick test results
Birth length | at baseline
  cm
Birth weight | at baseline
  g
anthropometrics | at baseline
  e.g. weight and lenght

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric hospital Bambino Gesù, Rome, Italy

IPD SHARING:
Plan to Share IPD: No